CLINICAL TRIAL: NCT05251714
Title: A Dose-confirming Study of CFI-402257 as a Single Agent in Advanced Solid Tumors and in Combination With Fulvestrant in Patients With ER+/HER2- Advanced Breast Cancer After Disease Progression on Prior CDK4/6 and Endocrine Therapy
Brief Title: CFI-402257, a Potent and Selective TTK Inhibitor, in Solid Tumors and With Fulvestrant in Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treadwell Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWT-203
Record Dates: First submitted 2022-02-07; First posted 2022-02-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Breast Cancer
Keywords: advanced solid tumors; advanced breast cancer; CFI-402257; 2257; fulvestrant; TWT-203; TWT203; UHN; University Health Network; Treadwell; Treadwell Therapeutics; endocrine therapy; TTK; TTK inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — CFI-402257; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion for monotherapy and combination arms with fulvestrant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Monotherapy Escalation and Expansion (Experimental): Dose selection and expansion of CFI-402257
  Interventions: Drug: CFI-402257
- Part B: Combination Escalation and Expansion (Experimental): Dose selection and expansion of CFI-402257 with Fulvestrant
  Interventions: Drug: CFI-402257; Drug: Fulvestrant

INTERVENTIONS:
Drug: CFI-402257 — Oral once daily in 28 day cycles
  Other Names: 2257; 402257
Drug: Fulvestrant — 500 mg given by IM injection on Day 1 and Day 15 of Cycle 1 and Day 1 of each subsequent cycle
  Other Names: Faslodex
  Arms: Part B: Combination Escalation and Expansion

SUMMARY:
The purpose of this study is to test the safety of an investigational drug called CFI-402257 alone in advanced solid tumors and in combination with Fulvestrant in advanced breast cancer patients.

DETAILED DESCRIPTION:
This study will be evaluating the safety and tolerability of CFI-402257 in subjects with advanced solid tumors and in advanced breast cancer. The study is designed to build on encouraging data from another study and to obtain further safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) data of CFI-402257.

ELIGIBILITY:
Inclusion Criteria: Part A Escalation

1. Have histological or cytological proof of advanced cancer that has progressed on at least 1 prior line of systemic therapy

Inclusion Criteria: Part A Expansion

1. Breast cancer patients positive for estrogen receptor and/or progesterone receptor and negative for HER2
2. Must have previously received a CDK4/6 inhibitor
3. No limit on lines of endocrine therapy
4. Must have received no more than 1 line of cytotoxic chemotherapy
5. Have measurable disease as per RECIST 1.1 guidelines.

Inclusion Criteria: Part B

1. Breast cancer patients positive for estrogen receptor and/or progesterone receptor and negative for HER2
2. Must have previously received a CDK4/6 inhibitor
3. Must have previously received no more than 1 line of endocrine therapy
4. Must have received no more than 1 line of cytotoxic chemotherapy
5. Have measurable disease as per RECIST 1.1 guidelines.

Exclusion Criteria: All Parts

1. Are pregnant or nursing.
2. Have received chemotherapy, biological therapy, or investigational treatment less than 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of study drug. Have received radiotherapy less than 2 weeks prior to first dose of study drug.
3. Received growth factors within 14 days prior to initiation of dosing of CFI-402257 or who will require ongoing treatment with growth factors
4. Have active, acute, or clinically significant chronic infections.
5. Have the following cardiovascular conditions

   * Have uncontrolled severe hypertension
   * Have symptomatic congestive heart failure
   * Have active angina pectoris or recent myocardial infarction
   * Have chronic atrial fibrillation or QTc of greater than 470 msec.
6. Have had major surgery within 21 days of starting therapy.
7. Primary central nervous system malignancies or known central nervous system metastasis.
8. Being treated with full dose warfarin.
9. Coagulopathy or any history of coagulopathy within the past 6 months, including history of deep vein thrombosis or pulmonary embolism.
10. Patients must avoid the use of strong CYP3A4 inducers and inhibitors. CYP3A sensitive substrates, PgP, BCRP inhibitors
11. Have had prior treatment with a TTK/MPS1 inhibitor.
12. Part B only: Known bleeding disorder which would prohibit administration of fulvestrant.
13. Part B only: Concomitant active malignancy other than ER+/HER2- advanced breast cancer.
14. Part A only: Concomitant active malignancy other than primary malignancy
15. Part B only: Had prior treatment with fulvestrant or agents with similar MoA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of adverse events of CFI-402257 as a single agent and at the recommended phase 2 dose (RP2D) | 48 months
  The number of subjects who experience an adverse event that was possibly related to study drug as assessed by CTCAE v 5.0.
To assess the incidence of adverse events of CFI-402257 in combination with fulvestrant and at the recommended phase 2 dose (RP2D) | 48 months
  The number of subjects who experience an adverse event that was possibly related to study drug as assessed by CTCAE v 5.0.

SECONDARY OUTCOMES:
Assessment of objective response rates | 48 months
  Objective response rate will be summarized by dose cohort and overall using the percent of patients in each tumor response category.
Assessment of objective response rates of the combination | 48 months
  Objective response rate will be summarized overall for advanced breast cancer patients
Assessment of the pharmacokinetic profile of CFI-402257 through AUC | 48 months
  Area under the plasma concentration (AUC) versus time curve from time 0 to time of least measurable concentration tabulated by dose group.
Assessment of the pharmacokinetic profile of CFI-402257 in combination with fulvestrant through AUC | 48 months
  Area under the plasma concentration (AUC) versus time curve from time 0 to time of least measurable concentration tabulated by dose group.
To evaluate the effect of CFI-402257 treatment on changes in variant allele function | 48 months
  Changes in variant allele function will be measured by looking at circulating tumor deoxyribonucleic acid compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: R Wesolowski, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - START San Antonio, San Antonio, Texas
  - START - Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialist, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
It is too early to determine whether we will make IPD available - we do not yet have a process written on this. Field will be updated once our policy / process is written.